CLINICAL TRIAL: NCT00267488
Title: An Open-label, Phase II, Multicenter Study of Intravenous Weekly Topotecan in Subjects With Recurrent or Persistent Endometrial Cancer
Brief Title: Intravenous Weekly Topotecan In Subjects With Recurrent Or Persistent Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100414
Record Dates: First submitted 2005-12-20; First posted 2005-12-21 (Estimated); Results first posted 2010-01-28 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-06

CONDITIONS: Neoplasms, Endometrial; Endometrial Cancer
Keywords: Hycamtin; endometrial cancer; topotecan
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: topotecan

SUMMARY:
The purpose of this study is to find out if Hycamtin given weekly is safe and effective for treating your endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* A subject will be eligible for inclusion in this study only if all of the following criteria are met:
* Subject has provided a written informed consent.
* Subject must be female and ≥18 years of age.
* Subjects' original endometrial carcinoma (any histologic type) must have had pathologic confirmation.
* Subject must have recurrent or persistent endometrial cancer.
* Subject must have at least one measurable lesion according to GOG-modified RECIST criteria.

  * Measurable disease must be accurately measured in at least one dimension (longest dimension to be recorded). Each lesion must be ≥ 20 mm when measured by conventional techniques, including palpation, plain X-ray, CT and MRI, or ≥10 mm when measured by spiral CT.
  * Measurable disease found on chest X-ray must be confirmed with CT or MRI. Either CT or MRI must be used throughout the study to further evaluate these lesions.
  * The same diagnostic method (CT, MRI, X-ray or physical exam) used to evaluate disease, must be used throughout the study to consistently evaluate lesions.
  * Palpable tumor masses that cannot be evaluated by CT or MRI scan should be evaluated by ultrasound or confirmed by biopsy.
  * Evaluable disease (measurable or non-measurable) may be in a field of prior radiation provided that at least six weeks have elapsed since receiving radiation and disease progression is clearly documented by radiographic study. It is preferential for the target lesion to be located outside an irradiated field.
  * Non-measurable disease is defined as all other lesions, including small lesions (longest diameter <20 mm with conventional techniques or <10 mm with spiral CT scan).
* Subject has received one prior chemotherapy regimen (excluding all topoisomerase I inhibitors e.g., HYCAMTIN and irinotecan).
* Subject is allowed to have received, but is not required to have received, one additional prior non-cytotoxic regimen for management of recurrent or persistent disease according to the following definition: Non-cytotoxic (biologic or cytostatic) agents include, but are not limited to, monoclonal antibodies, cytokines, and small molecule inhibitors of signal transduction. UM2004/00031/00 CONFIDENTIAL HCT100414 20
* Subject is at least 21 days from prior chemotherapy and at least 30 days from prior non-cytotoxic therapy and is recovered from associated toxicities.
* Subject must not have received radiotherapy for at least seven days.
* Subject must be at least three weeks since last major surgery (a lesser period is acceptable if deemed in the best interest of the subject). Subject must have an ECOG Performance Status of 0 or 1 (refer to
* Appendix 4, ECOG Performance Status).
* Subject must have, at screening, a probable life expectancy of at least three months.
* Subject of childbearing potential must be practicing adequate contraception [e.g., oral contraceptives, diaphragm plus spermicide, or intrauterine device (IUD)] or show documented complete abstinence from intercourse for at least three months prior to study start. The same contraceptive method should be used throughout the study and continue for at least four weeks after the end of the study. A subject will be considered of childbearing potential if not surgically sterile or post-menopausal (i.e., documented absence of menses for one year prior to entry into the study).

  14. Subject must have screening laboratory criteria as follows:
  * Hemoglobin ≥ 9.0 g/dL.
  * Neutrophils ≥ 1,500/mm³ [≥1.5 x 10^9/L].
  * Platelets ≥ 100,000/mm³ [≥100.0 x 10^9/L].
  * Creatinine ≤ upper limit of normal (ULN) or creatinine clearance (Clcreat) ≥ 60mL/min.
  * Creatinine clearance should be calculated using the Cockcroft-Gault formula:

Clcreat (mL/min) = (140-age [yr] x body wt [kg] x 0.85 72 x serum creatinine [mg/dL] OR Clcreat (mL/min) = 1.05 x (140-age [yr] x body wt [kg] serum creatinine [μmol/L]

* Serum bilirubin within normal limits.
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase < 2xULN if liver metastases are absent by abdominal CT or MRI or < 5xULN if liver metastases are present.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria are met:

* Subject is pregnant or lactating.
* Subject has received more than one prior chemotherapy regimen. UM2004/00031/00 CONFIDENTIAL HCT100414 21
* Subject has concomitant or history of previous malignancies, with the exception of adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer from which the subject has been disease-free for five years.
* Subject has active uncontrolled infection.
* Subject has brain metastases as documented by CT or MRI. Note: Asymptomatic subjects do not require CT or MRI to rule out brain metastases.
* Subject has received prior treatment with HYCAMTIN.
* Subject has a history of an allergic reaction to compounds chemically-related to HYCAMTIN or its constituents.
* Subject has received any investigational agent within 30 days or five half-lives (whichever is longer) prior to study entry.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2005-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (24):
- United States (19):
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Engelwood, Colorado
  - GSK Investigational Site, Coral Gables, Florida
  - GSK Investigational Site, Lakeland, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Hinsdale, Illinois
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Lincoln, Nebraska
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Chattanooga, Tennessee
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Seattle, Washington
- Canada (4):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
- GSK Investigational Site, Debrecen, Hungary

RESULTS

PARTICIPANT FLOW:
Groups:
- Topotecan Hydrochloride: Subjects received IV weekly Topotecan administered at either 2.5 mg/m2(if the subject had prior pelvic radiotherapy) or 3.0 mg/m2 on Days 1, 8 and 15(+ or - 2 days) every 28 days.
Period: Overall Study
Arm/Group | Topotecan Hydrochloride
Started | 37
Completed | 26
Not Completed | 11
Not completed — Sponsor Terminated Study | 9
Not completed — Protocol Violation | 1
Not completed — Other (Disease Progression) | 1

BASELINE CHARACTERISTICS:
Arm/Group | Topotecan Hydrochloride
Number analyzed (Participants) | 37
Age Continuous [Mean (Standard Deviation); unit: years] | 62.8 (9.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 34
  African Heritage/African American | 3

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response
Description: Tumor response based on GOG (Gynecological Oncology Group) modified RECIST (Response Evaluation Criteria In Solid Tumors) criteria. A 4-point scale used specifying tumor response. Complete Response (CR): Disappearance of all target lesions; Partial Response (PR): At least a 30% decrease in the sum of the LD of target lesions; (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD; (PD): At least a 20% increase in the sum of the LD of target lesions
Time Frame: Week 0 to Week 98 when endpoints were met
Population: Intent To Treat (ITT) Population - All subjects who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Topotecan Hydrochloride
Number analyzed (Participants) | 37
Participants
  Complete Response | 0
  Partial Response | 1
  Stable Disease | 9
  Progressive Disease | 23
  Unknown | 4

2. Secondary Outcome: Time to Progression
Description: Kaplan-Meier Estimate. Time to progression is defined as time from start of treatment until the first documented sign of disease progression or death due to progressive disease. Subjects who have not progressed or died at the time of analysis will be censored at the time of initiation of alternative anti-cancer therapy or time of last contact. Percentiles represent a set of points on a scale arrived at by dividing a group into parts in order of magnitude.
Time Frame: Week 0 to Week 19 when endpoints were met
Population: Intent To Treat (ITT) Population - All subjects who received at least one dose of study medication.
Measure: Mean (95% Confidence Interval); unit: Weeks
Arm/Group | Topotecan Hydrochloride
Number analyzed (Participants) | 37
Weeks
  25th percentile | 7.3 [6.9 to 8.1]
  Median percentile | 8.7 [7.9 to 11.1]
  75th percentile | 15.3 [9.0 to 19.1]

3. Secondary Outcome: Overall Survival
Description: Kaplan-Meier Estimate. Overall survival is defined as time from start of treatment until death due to any cause. Subjects who are alive at the time of analysis will be censored at the time of last contact.
Time Frame: Week 0 to Week 98
Population: Intent To Treat (ITT) Population - All subjects who received at least one dose of study medication.
Measure: Mean (95% Confidence Interval); unit: Weeks
Arm/Group | Topotecan Hydrochloride
Number analyzed (Participants) | 37
Weeks
  25th percentile | 20.4 [10.1 to 31.7]
  Median percentile | 47.3 [25.7 to 69.7]
  75th percentile | 89.3 [61.6 to 98.1]

4. Secondary Outcome: Response Duration
Description: The time from initial documented response to the first documented sign of progression or death due to progressive disease. Not calculated due to no Complete response and only 1 partial response.
Time Frame: Week 0 to week 98
Measure: Mean (95% Confidence Interval); unit: Weeks
Arm/Group | Topotecan Hydrochloride
Number analyzed (Participants) | 0

5. Secondary Outcome: Time to Response
Description: The time from start of treatment until the first documented response. Not calculated due to no Complete response and only 1 partial response.
Time Frame: Week 0 to week 98
Measure: Mean (95% Confidence Interval); unit: Hours
Arm/Group | Topotecan Hydrochloride
Number analyzed (Participants) | 0

6. Secondary Outcome: Safety and Tolerability as Summarized Through Adverse Event Reporting
Description: AE = Adverse Event reported at a frequency of greater than or equal to 16%. SAE = Serious Adverse Events where all were reported at 0% frequency.
Time Frame: Week 0 to week 98
Population: Intent To Treat (ITT) Population - All subjects who received at least one dose of study medication.
Measure: Number; unit: Number of Events
Arm/Group | Topotecan Hydrochloride
Number analyzed (Participants) | 37
Number of Events
  AE: Fatigue | 15
  AE: Nausea | 14
  AE: Constipation | 12
  AE: Abdominal Pain | 11
  AE: Vomiting | 8
  AE: Hypokalemia | 7
  AE: Anorexia | 6
  AE: Dyspnea | 6
  AE: Diarrhea | 6
  AE: Dizziness | 6
  AE: Headache | 6
  AE: Insomnia | 6
  SAE: Abdominal Pain | 2
  SAE: Gastrointestinal hemorrhage | 1
  SAE: Intestinal obstruction | 1
  SAE: Rectal Hemorrhage | 1
  SAE: Vomiting | 1
  SAE: Pulmonary Embolism | 3
  SAE: Dyspnea | 1
  SAE: Bacteremia | 1
  SAE: Streptococcal Bacteremia | 1
  SAE: Cerebral ischemia | 1
  SAE: Cerebral infarction | 1
  SAE: Incisional hernia, obstructive | 1
  SAE: Dehydration | 1
  SAE: Embolism venous | 1
  Alive at last contact-when follow-up ended | 9
  Deaths - any subject | 28
  Cause of Death - Disease of Study | 25
  Cause of Death - Non-Hematological toxicity | 2
  Cause of Death - Other-Brain Metastases | 1

ADVERSE EVENTS:
Arm/Group | Topotecan Hydrochloride
Serious Adverse Events (participants affected / at risk) | 11
Other Adverse Events (participants affected / at risk) | 34
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Topotecan Hydrochloride
Abdominal pain (Gastrointestinal disorders) | 2/37
Gastrointestinal hemorrahage (Gastrointestinal disorders) | 1/37
Intestinal Obstruction (Gastrointestinal disorders) | 1/37
Rectal hemorrhage (Gastrointestinal disorders) | 1/37
Vomiting (Gastrointestinal disorders) | 1/37
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3/37
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1/37
Bacteremia (Infections and infestations) | 1/37
Streptococcal Infection (Infections and infestations) | 1/37
Incisional hernia obstructive (Musculoskeletal and connective tissue disorders) | 1/37
Dehydration (General disorders) | 1/37
Embolism venous (Vascular disorders) | 1/37
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Topotecan Hydrochloride
Fatigue (General disorders) | 15/37
Nausea (Gastrointestinal disorders) | 14/37
Constipation (Gastrointestinal disorders) | 12/37
Abdominal pain (Gastrointestinal disorders) | 11/37
Vomiting (Gastrointestinal disorders) | 8/37
Hypokalemia (Metabolism and nutrition disorders) | 7/37
Anorexia (Metabolism and nutrition disorders) | 6/37
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6/37
Diarrhea (Gastrointestinal disorders) | 6/37
Dizziness (General disorders) | 6/37
Insomnia (Psychiatric disorders) | 6/37
Headache (Nervous system disorders) | 6/37
Back Pain (Musculoskeletal and connective tissue disorders) | 4/37
Cough (Respiratory, thoracic and mediastinal disorders) | 4/37
Hot Flush (General disorders) | 4/37
Pain (General disorders) | 4/37
Pharyngolanyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4/37
Arthralgia (Musculoskeletal and connective tissue disorders) | 3/37
Asthenia (Musculoskeletal and connective tissue disorders) | 3/37
Myalgia (Musculoskeletal and connective tissue disorders) | 3/37
Rectal Hemorrhage (Gastrointestinal disorders) | 3/37
Chest Pain (Cardiac disorders) | 3/37
Edema Peripheral (Vascular disorders) | 3/37
Dehydration (Metabolism and nutrition disorders) | 3/37
Hypomagnesaemia (Metabolism and nutrition disorders) | 3/37
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 3/37
Rash (Skin and subcutaneous tissue disorders) | 3/37
Urinary Tract infection (Renal and urinary disorders) | 3/37
Abdominal Distension (Gastrointestinal disorders) | 2/37
Blood Alkaline Phosphatase increased (Blood and lymphatic system disorders) | 2/37
Alopecia (Skin and subcutaneous tissue disorders) | 2/37
ALT increased (Hepatobiliary disorders) | 2/37
Anxiety (Nervous system disorders) | 2/37
Chills (General disorders) | 2/37
Dry Mouth (Gastrointestinal disorders) | 2/37
Hyponatraemia (Metabolism and nutrition disorders) | 2/37
Intestinal Obstruction (Gastrointestinal disorders) | 2/37
Blood Magnesium decreased (Metabolism and nutrition disorders) | 2/37
Pain in Extremity (General disorders) | 2/37
Pollakiuria (Renal and urinary disorders) | 2/37
Pyrexia (General disorders) | 2/37
Vaginal Discharge (Renal and urinary disorders) | 2/37
Weight Decrease (Metabolism and nutrition disorders) | 2/37

LIMITATIONS AND CAVEATS:
As there was only 1 responder, time to response, and duration of response were not calculated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.